CLINICAL TRIAL: NCT04611854
Title: Internet-delivered Therapy for Alcohol Misuse: Engagement, Outcomes and Satisfaction When Patients Select Preference for Self-guided or Guided Treatment
Brief Title: Internet-delivered Therapy for Alcohol Misuse: Investigating Patient Preference for Self-guided or Guided Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Centre for Patient-Oriented Research (Other); Saskatchewan Health Research Foundation (Other); Ministry of Health, Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-058b
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use Disorder
Keywords: Internet-delivered Cognitive Behaviour Therapy; Guidance; Alcohol Misuse
MeSH Terms: conditions — Alcoholism | interventions — Counseling; Ethanol

STUDY DESIGN:
Intervention Model Description: Each client will select either self-guided or guided option.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICBT for alcohol misuse: Guidance (Active Comparator): In this arm, participants will receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse with guidance from a health educator through regular weekly online messages. Participants may also be contacted through emails and phone calls. The team of guides consists of registered social workers, psychologists, and graduate students, with experience delivering ICBT.
  Interventions: Behavioral: Guidance; Behavioral: ICBT for alcohol misuse
- ICBT for alcohol misuse: Self-Guidance (Experimental): Participants who select this arm will receive the 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse. Participants are able to contact the Online Therapy Unit regarding any technical issues with logging onto the site. However, no guidance from a health educator will be provided. Clients will be monitored by providing brief measures on alcohol each week and measures of depression and anxiety administered at the beginning of week 5. However, clients will only be contacted if there is a significant clinical issue requiring attention (e.g., sudden increase in symptoms of depression and suicidal ideation).
  Interventions: Behavioral: ICBT for alcohol misuse

INTERVENTIONS:
Behavioral: Guidance — Guidance from a health educator through regular weekly online messages. Participants may also be contacted through emails and phone calls. The team of guides consists of registered social workers, psychologists, and graduate students, with experience delivering ICBT.
  Arms: ICBT for alcohol misuse: Guidance
Behavioral: ICBT for alcohol misuse — The 8-week internet-delivered cognitive behaviour therapy (ICBT) course for alcohol misuse. The course consists of 8 lessons distributed across 8 weeks.

SUMMARY:
Internet-delivered cognitive behaviour therapy (ICBT) shows promise as a method of treating alcohol misuse. In this form of treatment, patients complete online lessons over several weeks that assist patients in developing skills to address alcohol misuse. ICBT can be offered to patients in a self-guided format or with guidance. Self-guided ICBT allows users to complete lessons by themselves without any contact with a guide. Guided ICBT involves having support from a guide in the form of emails, online messages and/or brief telephone calls. In some studies, guided-ICBT has shown greater reductions in alcohol consumption than self-guided ICBT. To date, there has been limited research on patient preferences for these varying levels of support when ICBT is offered as part of routine health care. This represents an important research direction as there is some past research showing that patients' treatment preferences can affect study enrollment, attrition, adherence, satisfaction, and outcomes.

This study will investigate patient preferences for self-guided ICBT versus guided-ICBT and compare enrollment, attrition, adherence, and outcomes of the two approaches when patients select their treatment preferences. The study will also explore the extent to which preferences are related to patient background variables (e.g., duration, severity of problems, treatment goals in terms of patients wanting to cut-down on alcohol use versus to abstain from alcohol use). Furthermore, this study seeks to identify how ratings of effort and helpfulness throughout treatment vary depending on whether patients select self-guided versus guided ICBT. This study represents a pragmatic observational trial conducted in routine care and aims to increase understanding of how to implement ICBT within routine care.

ELIGIBILITY:
Inclusion Criteria:

* Timeline Followback (TLFB; preceding week alcohol consumption) > 13 drinks
* Alcohol Use Disorders Identification Test (AUDIT) > 7

Exclusion Criteria:

* Suicidal ideation (measured by scoring > 2 to question 9 of PHQ-9)
* Severe mental health or medical conditions
* Severe drug use problems (measured by scoring > 24 on Drug Use Disorders Identification Test [DUDIT] or clinical assessment)
* Low motivation to do, or concerns regarding, online treatment
* Ongoing or impending significant mental health treatment
* Not residing in Saskatchewan Canada for the duration of treatment
* Lack of or inconsistent access to a computer and internet at home or private place for the duration of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Drinks in preceding week as measured by Timeline Followback (TLFB) | Screening, Pre-treatment, 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment
  Change in preceding week alcohol consumption in terms of the total number of standard drinks consumed on each day during the previous 7 days.
Heavy drinking days preceding week as measured by Timeline Followback (TLFB) | Screening, Pre-treatment, 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment
  Change in preceding week alcohol consumption in terms of the total number of heavy drinking days during the previous 7 days.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Screening, 8 weeks (post-treatment), 3 months after treatment
  Change in alcohol-related problems and behaviours measured by total AUDIT score which can range from 0 to 40. Greater score indicates greater alcohol problems (worse outcome)
Penn Alcohol Craving Scale | Screening, 8 weeks (post-treatment), 3 months after treatment, 6 months after treatment, 12 months after treatment
  Change in alcohol craving as measured by a total score ranging between 0 to 30. Higher scores indicate greater craving (worse outcome).
Brief Situational Confidence Questionnaire (BSCQ) | Screening, 8 weeks (post-treatment), 3 months after treatment
  Change in confidence in resisting drinking urges in 8 situations rated from 0 to 100, rendering a sum score of 0-800. Higher scores indicate greater confidence (better outcome). There are 8 subscales, one for each item, assessed on a scale of 0-100. Thus, each subscale has a sum score of 0-100-. A higher score indicates greater confidence on the subscale.
Generalized Anxiety Disorder 7-item (GAD-7) | Screening, 8 weeks (post-treatment), 3 months after treatment
  Change in total GAD-7 anxiety score which can range from 0 to 21. Higher scores indicate greater anxiety (worse outcome).
Patient Health Questionnaire (PHQ-9) | Screening (Pre-treatment), 4 weeks (mid-treatment), 8 weeks (post-treatment), 3 months after treatment
  Change in total PHQ-9 score which can range from 0 to 27. Higher scores indicate greater depression (worse outcome).
Sheehan Disability Scale | Screening, 8 weeks (post-treatment), 3 months after treatment
  Change in three scores assessing functional impairment in three domains: 1) work/school, 2) social and 3) family life (each domain score ranges from 0 to 10, rendering a sum score of 0-30). Higher score indicates greater ability on the specified domain score (better outcome). Each domain score (subscale) renders a sum score of 0-10.
Treatment Credibility and Expectancy Scale | 4 weeks (mid-treatment)
  Measures the participant's thoughts and feelings about the treatment and the treatment's effectiveness in reducing participant's symptoms and increasing participant's functioning. Consists of 6 items. The first three of these and the 5th render a score of 1- 9. The other three questions render a score of 0-10. There are two subscales; 1) treatment credibility and 2) treatment expectancy. The first three questions are summed to render a score on the credibility subscale (0-27). The last three questions, the expectancy subscale, render a score of 0-29.
Readiness to Change Questionnaire Treatment Version (RCQ-TV) | Screening (Pre-treatment)
  Measures participants' motivation to change their drinking behaviours and determines at which stage of the Stages of Change model they are in (precontemplation, contemplation, or action). There is no sum score. Instead the items related to each stage are summed, and the individual is allocated to the stage that has the greatest score out of these three. (For more information about the scoring of this instrument, see Heather & Hönekopp, 2009).
Evaluation and Negative Effects Questionnaire | 8 weeks (post-treatment)
  This questionnaire will gather feedback from participants on perceived helpfulness and any negative effects experienced by participants during treatment. This brief questionnaire has been developed by the research team and does not have a sum score.
Lesson Completion | Ongoing throughout treatment (Weeks 1-8)
  The program website will record when patients access each lesson, providing a way to calculate the proportion of patients who complete each lesson and treatment overall.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Other researchers may ask to review IPD from this trial following completion of data collection. For the purposes of meta-analyses or other legitimate uses, IPD will be provided after being fully de-identified.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available for a period beginning 6 months after the conclusion of the trial until 5 years have elapsed.
Access Criteria: Data will be provided to researchers who provide a methodologically sound proposal and present a request for data that is within our operational capacity to provide. Additionally, researchers must provide information about how they will use and store the data, as well as sign an agreement related to the use of the data.

REFERENCES:
- [Derived] Sapkota RP, Lozinski T, Wilhems A, Nugent M, Schaub MP, Keough MT, Sundstrom C, Hadjistavropoulos HD. Internet-delivered therapy for alcohol misuse: engagement, satisfaction, and outcomes when patients select their preference for therapist- or self-guided treatment. Addict Sci Clin Pract. 2024 Apr 20;19(1):30. doi: 10.1186/s13722-024-00456-8. PMID 38643242